CLINICAL TRIAL: NCT03043963
Title: Mechanisms Underlying the Blood Pressure Lowering Effect of Sleep Extension
Brief Title: Mechanisms Underlying the Blood Pressure Lowering Effect of Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Janet M Mullington, PhD, Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015P000243
Record Dates: First submitted 2017-01-30; First posted 2017-02-06 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Timing (Active Comparator): Intervention will include basic education concerning sleep hygiene and regularity of sleep timing
  Interventions: Behavioral: Sleep Timing
- Sleep Extension (Experimental): Intervention will include basic education concerning sleep hygiene and an extension of the sleep period.
  Interventions: Behavioral: Sleep Extension

INTERVENTIONS:
Behavioral: Sleep Extension — Lengthen the duration of sleep time.
  Arms: Sleep Extension
Behavioral: Sleep Timing — Regularize the timing of the sleep period.
  Arms: Sleep Timing

SUMMARY:
The main purpose of this study is to learn about the influence of two different behavioral interventions (lasting 8 weeks) involving sleep for lowering blood pressure, and to study the mechanisms involved. There is research evidence that healthy sleep promotes heart-health and may decrease blood pressure, and that sensitivity to insufficient or disrupted sleep may be influenced by sex. This research will compare two interventions that are each designed to improve sleep health, and will investigate sex differences in response. The project includes 3 in-hospital stays with biological measurements to evaluate the underlying mechanisms associated with the effectiveness of two different blood pressure lowering behavioral interventions.

DETAILED DESCRIPTION:
The study involves home-based sleep-wake data collection before and during behavioral intervention, and 3 overnight stays in the hospital. For each hospital stay participants will be asked to arrive in the afternoon, and stay until the next evening. They will be provided dinner on the first day and breakfast, lunch and dinner on the second day. If they are taking any blood pressure medication they will continue to take it through the study. During the in-hospital stays, blood pressure will be measured continuously using two small finger cuffs. In order to monitor and record brain waves to determine sleep and wakefulness, small gold-coated disks called electrodes will be placed on the head and body. Heart rate, blood pressure and brain activity will be recorded for a little over 24 hours on each in-hospital stay. Before as well as during the in-hospital stays questions will be asked about sleep times, subjective sleepiness and other indices relating to well-being.

ELIGIBILITY:
Inclusion Criteria:

* pre-hypertension or stage one hypertension (BP ≥120/80 and <160/100).
* usual sleep period occurs at night

Exclusion Criteria:

* significant active or uncontrolled sleep disorders
* shiftwork
* current pregnancy
* diabetic patients who are insulin dependent (or have HbA1c>9.0%)
* current use of hypnotics or clonidine
* renal/electrolyte disorders and any other condition that the study screening physician considers would significantly impede participation in the study

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Reduction in 24 hour blood pressure | The primary outcome measure will be measured during 3 hospital visit periods of approximately 28 hours each. The primary outcome will be evaluated based on an 8 week behavioral intervention.
  24h blood pressure (daily averaged).

SECONDARY OUTCOMES:
Lowering of sleep period blood pressure | he primary outcome measure will be measured during 3 hospital visit periods ofThe secondary outcome will be evaluated based on an 8 week behavioral intervention.
  Blood pressure during day wake period minus blood pressure at night during sleep period

CONTACTS AND LOCATIONS:
Overall Officials: Janet M Mullington, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No